CLINICAL TRIAL: NCT05890651
Title: Holter and ECG Changes After Transcatheter Closure Of VSD In Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rasha Hassan Mahmoud, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Other Study IDs: soh-med-23-05-04MS
Record Dates: First submitted 2023-05-24; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: VSD Children
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG — Describe the electrocardiography (ECG) changes 24 hours,1,6,12 months after VSD transcatheter device closure in a pediatric population.

SUMMARY:
Ventricular septal defect (VSD) is the most common congenital heart now affecting children, which makes up 20 % of isolated congenital heart condition. Although VSD can develop in any area of the inter ventricular septum, the perimembranous VSD and muscular VSD which can occur anteriorly, posteriorly, inlet, or outlet, are the most frequent morphological forms. The supracristal varity is less prevelant.

While many VSDs close spontaneously, if they do not, large defects can lead to detrimental complications such as pulmonary arterial hypertension (PAH), ventricular dysfunction, and an increased risk of arrhythmias.

Hemodynamic impairment may arise according to the size and flow of the VSD. Hemodynamically unstable patients particularly benefit from a successful closure. After conventional open surgery to treat VSDs, complications from cardiopulmonary bypass, are infection, postpericardiotomy syndrome, chylothorax, and a full atrioventricular block are still conceivable (e.g., myocardial, and pulmonary injury, electrolyte imbalance, coagulopathy, and acute renal failure). Furthermore, when compared to nonsurgical treatments, prolonged postoperative stays in the ICU or hospital are required .

The requirements for transcatheter intervention are determined by the size and type of VSD. Transcatheter closure of a moderate-sized VSD with congestive heart failure, failure to thrive, substantially enlarged left atrium and LV, or increased pulmonary artery pressures is frequently recommended (or both). A pulmonary-to-systemic flow ratio larger than 2:1 is also required. Large VSDs with RV and pulmonary artery systolic pressures close to the left ventricular and aortic systolic pressures should be closed. Since the first case was reported in 1988 and had satisfactory results, catheter- based therapies have demonstrated promising results in comparison to surgery Arrhythmia, especially CAVB, is one of the most important complications after transcatheter occluder closure of pmVSD. The incident rate of arrhythmias in the early postoperative period ranges from 15.3% to 24.1% Bundle branch block was a common complication with the highest incident rate both in the early and long-term follow-up. During follow-up, nearly half of the conduction block could return to normal, some of which could be worse or even deteriorate into CAVB. Some of the reported late-onset CAVB cases have been observed with different degrees of conduction block in the early postoperative period.

Previous studies indicated that inlet occlusion increased the risk of LBBB whereas outlet occlusion decreased the associated risks.

the underlying mechanism of arrhythmias after transcatheter pmVSD closure is still unclear. The risk factors may include age, weight, operation duration time, operation technique, anatomy location of the pmVSD, size of the occluder, morphological characteristics of the occluder, and so on, but the conclusions about risk factor were different in various researches .

ELIGIBILITY:
Inclusion Criteria:

* All children under the age of 18 years diagnosed with VSD , that will undergo transcatheter VSD closure during the period of the study .

Exclusion Criteria:

* Failure to obtain informed consent .

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children under the age of 18 years diagnosed with VSD who will undergo transcatheter closure
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
ECG changes after VSD closure | 12 months
  the study will focus to describe the arrhythemia that occur after VSD closure also detect heart rate varibility a day before VSD closure and aday after closure detect long run arrythemia after VSD closure within one year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khoshhal SQ, Al-Mutairi MB, Alnajjar AA, Morsy MM, Salem SS, Al-Muhaya M, El-Harbi KM, Abo-Haded HM. Transcatheter device closure of ventricular septal defects in children: a retrospective study at a single cardiac center. Ann Saudi Med. 2020 Sep-Oct;40(5):396-402. doi: 10.5144/0256-4947.2020.396. Epub 2020 Oct 1. PMID 33007168
- [Background] Shah JH, Saraiya SP, Nikam TS, Jha MJ. Transcatheter Device Closure of Perimembranous Ventricular Septal Defect in Pediatric Patients: Long-Term Outcomes. Heart Views. 2020 Jan-Mar;21(1):17-21. doi: 10.4103/HEARTVIEWS.HEARTVIEWS_13_19. Epub 2020 Jan 23. PMID 32082495
- [Background] Li G, Liao H, Wu J, Zhou K, Hua Y, Wang C, Duan H, Shi X, Wu G, Li Y. Re-evaluation of the criteria for asymmetric amplatzer occluders in the closure of perimembranous ventricular septal defects: A case series report. Medicine (Baltimore). 2020 Aug 21;99(34):e21356. doi: 10.1097/MD.0000000000021356. PMID 32846756
- [Background] Mijangos-Vazquez R, El-Sisi A, Sandoval Jones JP, Garcia-Montes JA, Hernandez-Reyes R, Sobhy R, Abdelmassih A, Soliman MM, Ali S, Molina-Sanchez T, Zabal C. Transcatheter Closure of Perimembranous Ventricular Septal Defects Using Different Generations of Amplatzer Devices: Multicenter Experience. J Interv Cardiol. 2020 Feb 21;2020:8948249. doi: 10.1155/2020/8948249. eCollection 2020. PMID 32161516